CLINICAL TRIAL: NCT04184661
Title: Effect of Burosumab and 1-25 (OH) Vitamin D on Human Osteoclasts From Patients With Hypophosphatemic Rickets (HR)
Brief Title: Burosumab and 1-25 (OH) Vitamin D on Human Osteoclasts
Acronym: HYPO-CLASTE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0725; 2019-A02914-53 (Other: ID-RCB)
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hypophosphatemic Rickets
MeSH Terms: conditions — Rickets, Hypophosphatemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 25 mL blood sample will be collected on citrate tubes for osteoclastic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypophosphatemic rickets patients: 30 hypophosphatemic rickets patients older than 2 years will be included in this study
  Interventions: Other: blood sample
- controls patients: 10 controls patients from pediatric nephrology unit without hypophosphatemic rickets, older than 2 years will be included in this study
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 25 mL blood sample will be collected on citrate tubes for osteoclastic analysis.

SUMMARY:
Fibroblast growth factor 23 (FGF23) is the cornerstone of phosphate / calcium / vitamin D metabolism: it is synthesized mainly by osteocytes and acts as a Phosphating agent, inhibitor of dihydroxyvitamin D, and inhibitor of synthesis and secretion of Parathyroid hormone (PTH) in most tissues.

The specific role of FGF23 on bone has yet to be demonstrated. In some diseases such as hypophosphatemic rickets (HR), the direct role of FGF23 on bone has not yet been studied to our knowledge, whereas these genetic hypophosphatemias are secondary to overexpression of FGF23, whether an activating mutation of FGF23 or inhibitory mutations of its inhibitors (Dentin matrix acidic phosphoprotein 1 (DMP1) and Phosphate-regulating neutral endopeptidase, X-linked (PHEX)). However, patients with X-linked hypophosphatemic rickets (XLH) have higher circulating FGF23 levels than healthy controls and these levels are higher in treated patients.

Management of XLH consists primarily of correcting the native vitamin D defect by prescribing active vitamin D analogs as well as phosphate supplementation to improve bone mineralization and decrease dental complications, growth, and bone deformities. Recently, a new therapeutic option has been developed for XLH, burosumab, a human monoclonal antibody that binds and inhibits FGF23 activity. The use of burosumab is currently authorized in France in some pediatric patients with severe forms of XLH.

Independently of the indirect bone effects of phosphate correction and vitamin D levels, the direct role of burosumab on bone cells has never been studied. The objective of this project is to study the osteoclastic biology of patients with HR compared to control patients, and to evaluate the direct impact of the treatments used in this pathology on human osteoclasts.

ELIGIBILITY:
hypophosphatemic rickets patients:

Inclusion Criteria:

* children from 2 yars-old to 18 years old and adults
* patients with HR followed in the center of calcium and phosphorus metabolism rare diseases in Lyon-
* Patients and parent / holder of parental authority who have been informed of the study and do not object to participate

Exclusion Criteria:

* Patient being treated with oral corticosteroid or having received more than 3 months of corticosteroid treatment before surgery.
* Patients under tutorship or curatorship
* Pregnant and / or breastfeeding woman
* Patient deprived of liberty

Controls patients:

Inclusion Criteria:

* children from 2 years-old to 18 years old and adults
* patients with normal renal function (Schwartz glomerular filtration rate (GFR) >90 ml/min/1.73m²)
* Patients and parent / holder of parental authority who have been informed of the study and do not object to participate

Exclusion Criteria:

* Patient being treated with oral corticosteroid or having received more than 3 months of corticosteroid treatment before surgery.
* Patients under tutorship or curatorship
* Pregnant and / or breastfeeding woman
* Patient deprived of liberty
* Patient treated with immunosuppressive drugs
* Patient with inflammatory disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hypophosphatemic rickets and controls patients without hypophosphatemic rickets
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
number of osteoclastic cells obtained after at the end of differentiation | 1 day
  The analysis of osteoclastic differentiation will be obtained from the bone cells from patients with burosumab and/or 1-25 (OH) vitamin D

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Femme mère enfant, Bron
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Bicêtre Paris Saclay, Paris